CLINICAL TRIAL: NCT01210118
Title: The Effectiveness of High and Low Intensity Intervention for Smoking Cessation During Pregnancy
Brief Title: Interventions of Smoking Cessation During Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hellenic Anticancer Society (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, PANAGIOTIS BEHRAKIS, PROFESSOR OF NATIONAL AND KAPODISTRIAN UNIVERSITY OF ATHENS., Hellenic Anticancer Society
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBAL001
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Smoking Cessation
Keywords: Pregnancy; Smoking cessation; Cognitive-Behavioural interventions
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity intervention (Experimental): Experimental group participants received a higher intensity intervention, which include: 30 minutes of individualized cognitive-behavioural counselling delivered by a trained health care professional and a self-help manual especially tailored for smoking cessation during pregnancy. Counseling was based at the "5 Αs" (Ask,Advise, Asses, Assist, Arrange). In addition to counselling, a self help manual especially tailored for smoking cessation during pregnancy for Greek women was provided.
  Interventions: Behavioral: Higher intensity intervention
- Low intensity intervention (Other): Control group participants received a face to face low intensity intervention which lasted 5 minutes and included brief advice and the provision of a leaflet on smoking and pregnancy. This leaflet summarized the main effects of smoking during pregnancy and gave clear short messages for encouraging smoking cessation by setting up a quit date.
  Interventions: Behavioral: Low intensity intervention

INTERVENTIONS:
Behavioral: Low intensity intervention — Control group participants received a face to face low intensity intervention which lasted 5 minutes and included brief advice and the provision of a leaflet on smoking and pregnancy. This leaflet summarized the main effects of smoking during pregnancy and gave clear short messages for encouraging smoking cessation by setting up a quit date.
  Arms: Low intensity intervention
Behavioral: Higher intensity intervention — Experimental group participants received a higher intensity intervention, which include: 30 minutes of individualized cognitive-behavioural counselling delivered by a trained health care professional and a self-help manual especially tailored for smoking cessation during pregnancy. Counseling was based at the "5 Αs" (Ask,Advise, Asses, Assist, Arrange). In addition to counselling, a self help manual especially tailored for smoking cessation during pregnancy for Greek women was provided.
  Other Names: Experimental group
  Arms: High intensity intervention

SUMMARY:
The aim of this clinical trial is to test whether offering pregnant smokers a high intensity intervention for smoking cessation increases the rate of smoking cessation at the third trimester of pregnancy, compared to low intensity intervention for smoking cessation that is the usual care, control condition.

DETAILED DESCRIPTION:
This is a randomized controlled trial that compares the efficacy of a proactive pregnancy-tailored high intensity intervention for smoking cessation, with a usual care low intensity intervention, that is the control condition.

Intervention group participants will receive a high intensity intervention, which includes: 30 minutes of cognitive-behavioural intervention delivered by a trained health care professional through out the first 24 weeks of gestation and a self-help manual especially tailored for smoking cessation during pregnancy. Control group participants will receive 5 minutes of low intensity intervention.

Participants' smoking status will be biochemically validated with urine cotinine and nicotine both at the baseline and at the 32nd week of gestation, expired carbon monoxide (CO) will be measured only at the baseline. After childbirth the infants' birth weight, the premature birth and any other complications in pregnancy and childbirth will be recorded. No medication is going to be used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* current cigarette smoker (smoked >5 cigarettes in the past 7 days)
* 18 years old or older

Exclusion Criteria:

* More than 24 weeks' gestation at study entry
* No telephone access
* Not planning to live in Athens for 1 year
* Unable to read and speak Greek
* Alcoholics
* Use of drug substances
* Depression

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis K Behrakis, Professor, Study Chair — National and Kapodistrian University of Athens; Andriani N Loukopoulou, PhD pending, Principal Investigator — National and Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Peripheral General Hospital-Maternity Helena Venizelos, Athens, Attica
  - Maternity Unit of ATTIKON University Hospital, Haidari, Attica

REFERENCES:
- [Background] Loukopoulou A N, Evangelopoulou V, Behrakis P K.Smoking and pregnancy. Pneumon 23(2):160-167,2010.
- [Background] Loukopoulou AN, Vasiliou MP, Behrakis PK. (2011) Interventions for smoking cessation during Pregnancy Pneumon, 24(1):381-391(Review).
- [Background] Loukopoulou AN, Vardavas CI, Farmakides G, Rossolymos C, Chrelias C, Tzatzarakis MN, Tsatsakis A, Lymberi M, Connolly GN, Behrakis PK. Design and study protocol of the maternal smoking cessation during pregnancy study, (M-SCOPE). BMC Public Health. 2011 Dec 6;11:903. doi: 10.1186/1471-2458-11-903. PMID 22145828
- [Derived] Loukopoulou AN, Vardavas CI, Farmakides G, Rosolymos C, Chrelias C, Tzatzarakis M, Tsatsakis A, Myridakis A, Lyberi M, Behrakis PK. Counselling for smoking cessation during pregnancy reduces tobacco-specific nitrosamine (NNAL) concentrations: A randomized controlled trial. Eur J Midwifery. 2018 Nov 14;2:14. doi: 10.18332/ejm/99546. eCollection 2018. PMID 33537575
- See also: MedlinePlus related topics: Pregnancy, Smoking Cessation — http://www.nlm.nih.gov/medlineplus/quittingsmoking.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research took place in two hospitals situated in the area of Attici, Greece namely through the Peripheral General Maternity Hospital 'Helena Venizelos' and the Maternity Unit of the 'Attikon' University Hospital. Recruitment lasted from November 2009- February 2011.
Pre-assignment Details: Sixty-six enrolled participants were excluded from the trial before assignment to groups because 36 of them did not meet the inclusion criteria and 30 of them refused to participate.
Groups:
- High Intensity Intervention: Experimental group participants received a higher intensity intervention, which included: 30 minutes of individualized cognitive-behavioural counselling delivered by a trained health care professional and a self-help manual especially tailored for smoking cessation during pregnancy. Counseling was based at the "5 Αs" (Ask,Advise, Asses, Assist, Arrange). In addition to counselling, a self help manual especially tailored for smoking cessation during pregnancy for Greek women was provided.
Period: Overall Study
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Started | 45 | 47
Completed | 42 | 42
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Spontaneous abortion | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity Intervention | Low Intensity Intervention | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.9) | 32.4 (4.5) | 31.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Participants' Smoking Status
Description: participants' smoking status was validated by urine cotinine and urine nicotine
Time Frame: around the 32nd week of gestation.
Population: Only the participants who met the inclusion criteria and completed the research protocol were included in the research analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Number analyzed (Participants) | 42 | 42
ng/ml
  Urine nicotine | 253.6 (532.3) | 678.9 (1467.2)
  Urine cotinine | 311.9 (490.1) | 479.6 (563.4)

2. Secondary Outcome: Birth Weight
Description: Infants' birth weight was recorded.
Time Frame: After child birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: birth weight in grams
Groups:
- High Intensity Intervention: Experimental group participants received a higher intensity intervention, which include: 30 minutes of individualized cognitive-behavioural counselling delivered by a trained health care professional and a self-help manual especially tailored for smoking cessation during pregnancy. Counseling was based at the
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Number analyzed (Participants) | 42 | 42
birth weight in grams | 3,003.4 (499.8) | 3,231.3 (450.8)

3. Primary Outcome: The Effectiveness of the Interventions According the Levels of Urine Cotinine Before and After Intervention.
Description: The basic primary outcomes of the study present the levels of urine cotinine before and after intervention separately for each group according to the cut of point that is used for the separation of active from passive smoking ,when urine cotinine ≤80ng/ml: there is biochemically validated smoking cessation.
Time Frame: At the baseline and at the 32nd week of gestation
Measure: Number; unit: percentage of participants who quit
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Number analyzed (Participants) | 42 | 42
percentage of participants who quit
  Before Intervention (baseline) | 11.9 [0.001 to 0.001] | 21.4 [0.001 to 1.000]
  After intervention (32nd week of gestation) | 45.2 | 21.4

4. Secondary Outcome: Days of Prematurity of Birth
Description: Days of prematurity of birth were recorded
Time Frame: After child birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of days
Groups:
- High Intensity Intervention: Experimental group participants received a higher intensity intervention, which included: 30 minutes of individualized cognitive-behavioural counselling delivered by a trained health care professional and a self-help manual especially tailored for smoking cessation during pregnancy. Counseling was based at the
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Number analyzed (Participants) | 42 | 42
number of days | 14.3 (11.6) | 10.5 (6.9)

ADVERSE EVENTS:
Arm/Group | High Intensity Intervention | Low Intensity Intervention
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No